CLINICAL TRIAL: NCT00774748
Title: Once Weekly Subcutaneous Ports for the Administration of Anticoagulants - A Prospective Pharmacokinetic and Clinical Utilization Study
Brief Title: Once Weekly Subcutaneous Ports for the Administration of Anticoagulants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: IntraPump Infusion Systems (Industry); Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Insuflon07-1631
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2012-01

CONDITIONS: Venous Thromboembolism
Keywords: low molecular weight heparin; enoxaparin; Lovenox; Insuflon; subcutaneous catheter; once or twice daily dosing of subcutaneous enoxaparin
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): All participants in the study will use the subcutaneous catheter twice for a period of one week each to inject the enoxaparin. For the remainder of the study the participants will inject subcutaneously.
  Interventions: Device: Insuflon

INTERVENTIONS:
Device: Insuflon — Indwelling subcutaneous catheter indicated for subcutaneous infusion of medication by injection. Maximum lifespan: 7 days or 75 injections.
  Other Names: Insuflon catheter; device number K881767

SUMMARY:
The purpose of this study is to ascertain whether subcutaneous ports are an effective and reliable way to administer the low molecular weight heparin (LMWH) enoxaparin to patients for the prevention or treatment of venous thromboembolism.

DETAILED DESCRIPTION:
Subcutaneous ports have recently been used to administer Low Molecular Weight Heparin (LMWH) to patients for the prevention or treatment of venous thromboembolism; however, no studies have been performed to evaluate the ports' reliability in delivering this type of drug. Hence, it is not known whether absorption of the drug is constant over the seven-day lifespan of the port. Although the use of subcutaneous ports is not currently the standard of care, health care providers are more frequently using this as an alternative method to direct injection of LMWH, particularly in pediatric patients.

The main advantage of subcutaneous ports is the decreased number of needle sticks when using the ports to administer the medication. However, it is possible that, due to potential repeated bleeding into the subcutaneous space at the port site or other factors, drug absorption may decrease over the seven day lifespan of the port, resulting in a decrease of plasma drug level. Subtherapeutic LMWH levels and, hence, ineffective anticoagulation may result. This study's aim is to determine if the current use of subcutaneous ports is a safe, effective and reliable way of administering LMWH for the purpose of anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving once or twice daily dosing of therapeutic doses of subcutaneous Enoxaparin.
* Subject has been on the same dose of Enoxaparin for at least one week.
* Anticipated length of Enoxaparin treatment at least 4 weeks.
* Age ≥ 18 years.
* Subject demonstration of proper subcutaneous catheter care during one education session with the investigator.

Exclusion Criteria:

* Chronic renal insufficiency with glomerular filtration rate < 30 mL/min.
* Pregnancy
* Venous thromboembolism within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Moll, MD, Principal Investigator — University of North Carolina at Chapel Hill School of Medicine Department of Medicine
Locations (1):
- University of North Carolina at Chapel Hill School of Medicine; University of North Carolina Hospital, N.C. Memorial Hospital, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insuflon: All participants in the study will use the subcutaneous catheter twice for a period of one week each to inject the enoxaparin. For the remainder of the study the participants will inject subcutaneously.
Period: Overall Study
Arm/Group | Insuflon
Started | 21
Completed | 18
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Insuflon
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Secondary Outcome: Percent Difference of Each Participant's Subcutaneous Anti-Xa Levels
Description: Anti-Xa subcutaneous blood levels are displayed in percent difference to show normal fluctuations of anti-Xa levels without using the port. A percent difference is calculated by the current value has the previous value subtracted from it; this new number is divided by the absolute value of the previous value; then this new number is multiplied by 100. This allows each set of data to be compared to itself. Anti-Xa tests measure the concentration of low molecular weight heparin in the blood.
Time Frame: 6 time points (for each participant) in approximately 3 months
Population: All participants were represented with a baseline fluctuation in percent difference.
Measure: Median (Full Range); unit: Percent
Groups:
- All Participants: Both dosing schedules, once and twice daily, all participants.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Percent | 12 [1.4 to 35.6]

2. Secondary Outcome: Percent Difference of Each Participant's Anti-Xa Levels Without Port and Day One of Using the Port
Description: Comparing subcutaneous baseline (without port) anti-Xa levels with day one of using the port. A percent difference is calculated by the current value has the previous value subtracted from it; this new number is divided by the absolute value of the previous value; then this new number is multiplied by 100. This allows each set of data to be compared to itself. Anti-Xa tests measure the concentration of low molecular weight heparin in the blood.
Time Frame: approximately 3 months
Population: Twenty participants, excluding one outlier of 97%.
Measure: Median (Full Range); unit: Percent
Groups:
- All Participants: All participants on both dosing schedules, once and twice daily LMWH.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Percent | 14 [0 to 68]

3. Secondary Outcome: Percent Difference of Each Participant's Anti-Xa Blood Levels Between Day 1 and Day 7
Description: Comparing anti-Xa levels from the first day of using the port and the last day of using the port. A percent difference is calculated by the current value has the previous value subtracted from it; this new number is divided by the absolute value of the previous value; then this new number is multiplied by 100. This allows each set of data to be compared to itself. Anti-Xa tests measure the concentration of low molecular weight heparin in the blood.
Time Frame: 7 days
Population: All participants, excluding two outliers of 97% and 150%
Measure: Median (Full Range); unit: Percent
Groups:
- All Participants: All participants on both dosing schedules, once and twice daily.
Arm/Group | All Participants
Number analyzed (Participants) | 17
Percent | 16 [1.5 to 65]

4. Primary Outcome: Average Subcutaneous Anti-Xa Blood Levels
Description: Blood levels taken from the first and last visits (when available) were combined to get an average. The anti-Xa test reports the low molecular weight heparin concentration in the blood.
Time Frame: approximately 3 months
Population: Participants were separated into the two dosing schedules, since the target anti-Xa level is different for the two different types of doses. The once daily dosing sub-group was analyzed for this primary outcome measure.
Measure: Mean (Full Range); unit: IU/mL
Groups:
- Once Daily Dosing: 10 participants were placed on an once daily dosing schedule in accordance with their physician approved, standard of care weight specific dosage.
Arm/Group | Once Daily Dosing
Number analyzed (Participants) | 10
IU/mL | 1.43 [1.41 to 1.56]

5. Secondary Outcome: Standard Deviation of Participant's Own Glomerular Filtration Rate (GFR)
Description: GFR was calculated from a creatinine blood level to establish a safe renal function that would validate anti-Xa levels. Low molecular weight heparin is primarily cleared from the body by the kidneys. Any condition that decreases kidney function can potentially decrease LMWH clearance, increasing its concentration in the blood and increasing the potential for excessive bleeding.
Time Frame: 6 time points in approximately 3 months
Population: Included all participants who had at lease one visit and one blood draw.
Measure: Mean (Full Range); unit: mL/min
Groups:
- All Participants: All participants on both a daily and twice daily dosing schedule
Arm/Group | All Participants
Number analyzed (Participants) | 21
mL/min | 6.75 [0 to 13.5]

ADVERSE EVENTS:
Arm/Group | Insuflon
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insuflon (N=21)
Subject had a recurrent deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1) — Recurrent blood clots are a risk for patients who have already had a clot. This event was not related to the study procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No